CLINICAL TRIAL: NCT01959308
Title: Adherence to Immunosuppressive Therapy in Adult and Adolescent Liver Transplant Recipients: A Questionnaire Survey
Brief Title: Adherence to Immunosuppressive Therapy Liver Transplant Recipients
Acronym: AIM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: AIM Study
Record Dates: First submitted 2013-10-08; First posted 2013-10-10 (Estimated); Last update posted 2013-10-10 (Estimated); Status verified 2013-10

CONDITIONS: Focus : To Study the Differences in Patient Compliance to Immunosuppressive Treatments and Patient Preference.
Keywords: Adherence; Compliance; Immunosuppressive Therapy; Liver Transplant; Liver Recipients; Adult; Adolescent
MeSH Terms: conditions — Patient Preference; Patient Compliance

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Immunosuppressive therapy: Liver Transplant recipients who are receiving various doses and types of immunosuppressive therapy

INTERVENTIONS:
Other:

SUMMARY:
Immunosuppressive therapy is fundamental in post-liver transplant patients to prevent and reduce the incidence of acute cellular rejection. Non-compliance to treatment leading to graft rejection is a well-recognized event. This study aims to study the differences in patient compliance to immunosuppressive treatments and patient preference.

DETAILED DESCRIPTION:
Patient's demographic details such as age, gender, body mass index, education level, language, and occupation will be captured. Clinical details such as significant comorbidities, date of liver transplant, type of transplant (cadaveric or living related), underlying liver disease, type of immunosuppressants, and history of rejection with its details will also be recorded.

Participants will be asked to fill in a Questionnaire aimed to capture socioeconomic and clinical background, as well as the number, type, and dosing schedule of their immunosuppressants. Details and frequency of missed doses, the reason for 'missed doses', and patient's dosing preferences will be the questionnaire to access patient's compliance to medication. A liver transplant coordinator trained to administer the questionnaire will assist patients if required.

The participant will be approached either during their clinic visit or through phone call. For participants who are approached during their clinic session, informed consent process will be conducted in the clinic by the assigned study team member(s). Participants will then complete the questionnaire. Some participants may be on 6-monthly or annual follow-up. For this group of participants, a phone call will be made to ask if they would be keen to participate in this questionnaire study. If they are agreeable, 2 copies of DSRB approved version of informed consent forms together with the questionnaire form will be posted to participants for their completion. Participant will sign the informed consent forms, complete the questionnaire and post the completed documents back to study team members.

The primary and secondary outcome is patient compliance and patient preference, respectively. Besides the type of immunosuppressants, factors associated with outcomes will also be analyzed. Data entry and analysis will be conducted using SAS 9.2. Differences in categorical variables will be analyzed with chi-square test and Fisher's-exact test where appropriate and differences in continuous variables will be analyzed with student T-test. A two-sided analysis will be used and a p value of <0.5 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, 18 years old and above
* Written informed consent must be obtained from subjects prior to study participation

Exclusion Criteria:

* Patients who have not received any immunosuppresants post liver transplant surgery
* Patients who are not willing to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients (males or females age 18 years and above) who are on active follow up at liver transplant clinic at National University Hospital, Singapore.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-06; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Compliance / Adherence to immunosuppression | 1 year
  1. Determine compliance to immunosuppressive therapy among liver transplant patients followed up in Liver Transplant Clinic in NUH
  2. Elucidate factors associated with their compliance level

SECONDARY OUTCOMES:
Patient preferences on dosing of immunosuppression & associated factors | 1 year
  1. Determine their preferences on the dosing frequency of immunosuppressive administration
  2. Elucidate factors associated with their preferences.

CONTACTS AND LOCATIONS:
Locations (1):
- National University Hospital, Div of Gastroenterology & Hepatology, National University Center for Organ Transplantation, Singapore, Singapore